CLINICAL TRIAL: NCT00968175
Title: EUS Guided-Celiac Plexus Neurolysis (CPN) for Patients With Unresectable Pancreatic Cancer: A Multi-Center, Randomized, Single-Blinded Controlled Trial
Brief Title: Endoscopic Ultrasound (EUS) Guided-Celiac Plexus Neurolysis (CPN) in Unresectable Pancreatic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: AdventHealth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: F090528002
Record Dates: First submitted 2009-08-26; First posted 2009-08-28 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-05

CONDITIONS: Pain; Pancreatic Cancer
Keywords: Ultrasound guided celiac plexus neurolysis; CPN; Pancreatic Cancer; Pain Management
MeSH Terms: conditions — Pain; Pancreatic Neoplasms; Agnosia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1: CPN + analgesic therapy (Active Comparator): Receives ultrasound guided celiac plexus neurolysis (CPN) in addition to standard analgesic therapy
  Interventions: Procedure: Ultrasound guided celiac plexus neurolysis (CPN)
- Analgesic therapy alone (No Intervention): Will not receive ultrasound guided celiac plexus neurolysis (CPN); only standard analgesic therapy for pain management

INTERVENTIONS:
Procedure: Ultrasound guided celiac plexus neurolysis (CPN) — Initial procedure and rescue procedure if applicable
  Other Names: EUS-CPN
  Arms: Group 1: CPN + analgesic therapy

SUMMARY:
The purpose of this study is to examine endoscopic ultrasound guided celiac plexus neurolysis (CPN) with analgesic therapy in patients with unresectable pancreatic cancer as it applies to decreasing the severity of abdominal pain when compared to analgesic therapy alone.

DETAILED DESCRIPTION:
The specific primary aim of this study is to evaluate the efficacy of EUS-CPN + analgesic therapy (Group 1) in pain relief of patients with unresectable pancreatic cancer when compared with analgesic therapy (Group 2). The hypothesis will be tested by comparing the changes in reported pain severity between those who receive EUS-CPN in addition to analgesic therapy as compared to analgesic therapy alone.

The secondary aims of this study are to evaluate the efficacy of EUS-CPN + analgesic therapy in improvement of quality of life (QOL) of patients with unresectable pancreatic cancer when compared to when compared with analgesic therapy alone, compare pain medication usage between Group 1 when compared to Group 2, and compare the referral for rescue block during the course of the study between Group 1 and Group 2

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female
2. Age ≥19 yrs old
3. Abdominal pain typical for pancreatic cancer ≥3/10
4. Abdominal CT radiologically consistent with the diagnosis of pancreatic cancer
5. Pancreatic cancer confirmed by FNA during EUS
6. Inoperability of pancreatic cancer as determined during EUS or prior CT

Exclusion Criteria:

1. Age < 19 yrs old
2. Unable to safely undergo EUS for any reason
3. Coagulopathy (prolongation of prothrombin time > 18 sec, thrombocytopenia <80,000 platelets/ml)
4. Previous CPN or other neurolytic block that could affect pancreatic cancer -related pain or had implanted epidural or intrathecal analgesic therapy
5. Another cause for abdominal pain such as pseudocyst, ulcer or other intra-abdominal disorder
6. Potential patient noncompliance (refusing to follow schedule of events)
7. Active alcohol or other drug use or significant psychiatric illness
8. Pregnant or breastfeeding
9. Unable to consent
10. Non-English speaking

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-06; Primary Completion 2013-03 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The efficacy of EUS-CPN and analgesic therapy in pain relief of patients with unresectable pancreatic cancer when compared with analgesic therapy | ~ 2 year

SECONDARY OUTCOMES:
To evaluate the efficacy of EUS-CPN and analgesic therapy in improvement of quality of life (QOL) | ~2 year

CONTACTS AND LOCATIONS:
Overall Officials: Jayapal Ramesh, MD, Principal Investigator — University of Alabama at Birmingham
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Florida Hospital, Orlando, Florida